CLINICAL TRIAL: NCT04521751
Title: Lean Efficacy Phase IIa Proof of Concept Trial (LEAAP). A Study in Overweight and Obese Patients During Twenty-six Weeks, Investigating the Effect of EMP16-02 on Body Weight, Safety and Clinical Biomarkers
Brief Title: A Proof of Concept Trial in Overweight and Obese Patients, Investigating Effect of EMP16-02 on Body Weight (Primary)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Empros Pharma AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EP-002
Record Dates: First submitted 2020-05-14; First posted 2020-08-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2021-08

CONDITIONS: Overweight or Obesity
Keywords: Overweight; Obesity; Orlistat; Acarbose
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This is an exploratory, randomised, double-blind and placebo-controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study and the allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.
  Active treatment and placebo capsules are identical in appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMP16-02 120 mg orlistat/40 mg acarbose (Experimental): Dosage form: Oral, modified-release (MR) fixed dose combination (FDC) of orlistat and acarbose formulated in capsules.
  Dosage: 120 mg O/40 mg A (given as 2 capsules EMP16-02-60/20). Frequency: Three times daily (TID) together with the three main daily meals .Taken halfway through each meal, together with approximately 100-200 mL water (or other drink).
  Duration: 26 weeks.
  Interventions: Drug: EMP16-02 120 mg orlistat/40 mg acarbose
- EMP16-02 150 mg orlistat/50 mg acarbose (Experimental): Dosage form: Oral, modified-release (MR) fixed dose combination (FDC) of orlistat and acarbose formulated in capsules.
  Dosage: 150 mg O/50 mg A (given as 1 capsule EMP16-02-90/30 and 1 capsule EMP16-02-60/20).
  Frequency: Three times daily (TID) together with the three main daily meals .Taken halfway through each meal, together with approximately 100-200 mL water (or other drink).
  Duration: 26 weeks.
  Interventions: Drug: EMP16-02 150 mg orlistat/50 mg acarbose
- Placebo (Placebo Comparator): Dosage form: Matching, oral capsule. Identical in appearance but contain only cellulose.
  Dosage: Placebo (given as 2 placebo capsules) Frequency: Three times daily (TID) together with the three main daily meals .Taken halfway through each meal, together with approximately 100-200 mL water (or other drink).
  Duration: 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMP16-02 120 mg orlistat/40 mg acarbose — EMP16-02 capsules are composed of three pharmaceutical fractions (granules denoted G1, G2 and G3). G1= Prolonged release of acarbose, G2= Enteric-coated granule fraction containing orlistat and acarbose, G3= Orlistat with a delayed on-set release mechanism.
  Other Names: 120 mg O/40 mg A
  Arms: EMP16-02 120 mg orlistat/40 mg acarbose
Drug: EMP16-02 150 mg orlistat/50 mg acarbose — EMP16-02 capsules are composed of three pharmaceutical fractions (granules denoted G1, G2 and G3). G1= Prolonged release of acarbose, G2= Enteric-coated granule fraction containing orlistat and acarbose, G3= Orlistat with a delayed on-set release mechanism.
  Other Names: 150 mg O/50 mg A
  Arms: EMP16-02 150 mg orlistat/50 mg acarbose
Drug: Placebo — Matching oral placebo capsules
  Arms: Placebo

SUMMARY:
This study is a proof of concept study to demonstrate that EMP16-02, a fixed dose combination (FDC) of orlistat and acarbose in an oral multiple-unit modified release (MR) formulation leads to a clinically relevant decrease in body weight. The study aims to evaluate the efficacy, safety and tolerability of treatment with two different doses of EMP16 02 (120 mg orlistat/40 mg acarbose and 150 mg orlistat/50 mg acarbose) for 26 weeks on reducing body weight in obese patients.

DETAILED DESCRIPTION:
This study is a proof of concept study to demonstrate that EMP16-02, a fixed dose combination (FDC) of orlistat and acarbose in an oral multiple-unit modified release (MR) formulation leads to a clinically relevant decrease in body weight. The study aims to evaluate the efficacy, safety and tolerability of treatment with two different doses of EMP16 02 (120 mg orlistat/40 mg acarbose and 150 mg orlistat/50 mg acarbose) for 26 weeks on reducing body weight in obese patients.

EMP16-02 will be given to obese patients with an initial BMI ≥ 30 kg/m² or ≥ 28 kg/m² in the presence of other risk factors (e.g., hypertension, glucose dysregulation such as impaired glucose tolerance and type 2 diabetes mellitus (T2DM) and/or dyslipidaemia.

The study consists of 6 visits to the research clinic, including screening and follow-up. There will be no overnight stays at the clinic.

Visit 1: Screening (Visit 1) will take place from Day -28 to Day -1. Visit 2: Eligible and consenting patients will arrive at the research clinic in the morning of the first dosing day (Day 1, Visit 2) after at least 8 hours overnight fasting.

A re-check of eligibility including a brief physical examination, vital signs and assessment of body weight will be conducted. The patients will be randomised to either of two doses of EMP16-02 or placebo:

1. EMP16-02 120 mg O/40 mg A
2. EMP16-02 150 mg O/50 mg A
3. Placebo (identical capsules) Blood sampling (fasting), and anthropometric measurements will be performed. Patients will receive electronic diary instructions and will be asked to fill in a satiety and craving questionnaire before breakfast (at the clinic), and then once every hour for 4 hours until before lunch (at home). A standardised breakfast will be served at the clinic. Halfway through breakfast at Visit 2, all patients will receive a placebo capsule independent of the treatment arm to which the patients have been randomised, to provide patients with the opportunity to train on self administering the Investigational Medicinal Product (IMP) under supervision of clinic staff. The patients will also receive instructions for filling in more questionnaires regarding health and quality of life, meal pattern, activity and sleep, and gastrointestinal symptoms (gastrointestinal rating scale [GSRS]). The patients will be instructed to take EMP16-02 or placebo halfway through each meal, together with approximately 100-200 mL water (or other drink) on all subsequent treatment days. Once IMP has been handed out, the patients are free to leave the clinic. The first randomised IMP dose will be taken during lunch (or the next meal) at home.

Between visit 2 and 3: Patients randomised to EMP16-02 will start with a run-in period of 6 weeks during which the dose is sequentially increased. From week 7, all patients will have reached their final intended dose and a 20 week treatment and observation period will start. The run-in phase will start at a dose of 60 mg O and 20 mg A TID, which will sequentially be increased with 30 mg O/10 mg A every two weeks until the target doses of 120 mg O/40 mg A TID (for the lower dose group) and 150 mg O/50 mg A TID (for the higher dose group) are reached. Placebo treatment consists of matching oral capsules. Placebo and EMP16-02 capsules need to be taken TID together with three daily meals.

Visit 3-5: Patients will come to the clinic at Visit 3 (week 7), Visit 4 (week 14) and Visit 5 (week 26) for safety assessments and assessments of weight and anthropometric measurements. Patients will arrive in the morning after at least 8 hours overnight fasting. All visits will start with a brief physical examination followed by blood sampling (fasting) and assessment of body weight and body composition. A standardised breakfast will be served during which the patient will take the IMP. All or a selection of the questionnaires, including the satiety and craving questionnaire, will be filled in in a similar way as during Visit 2.

New IMP will be handed out to the patients at Visit 2, 3 and 4. At Visit 5 (week 26), the patients will take the last dose during breakfast at the clinic.

After 18 and 22 weeks of treatment (Day 123 ± 3 days and Day 151 ± 3 days, respectively), patients will be asked to answer questions about IMP compliance, occurrence of adverse events (AEs) and use of concomitant medication using an electronic diary.

Visit 6: A follow up safety visit.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Aged ≥ 18 and ≤ 75 years.
3. BMI ≥ 30 or ≥ 28 kg/m² in the presence of other risk factors based on patient interview, e.g., hypertension (either or not treated with antihypertensive agents), glucose dysregulation such as impaired glucose tolerance (defined as elevated fasting glucose or HbA1c as judged by the Investigator) and T2DM that is treated with life style changes (no medication allowed), and/or dyslipidaemia (either or not treated with antihyperlipidemic agents). If indicated, plasma/serum total cholesterol, LDL, HDL, and triglycerides can be measured to verify eligibility as judged by the Investigator.
4. Acceptable medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
5. Adequate renal and hepatic function as judged by the Investigator in accordance with the expected disease profile
6. Weight stable (<5% reported change during the three months preceding screening), based on patient interview and weight assessments at screening (Visit 1) and randomisation (Visit 2).
7. Willing to eat three meals per day, and willing to eat breakfast during the visits to the clinic.
8. Males and females may be included in the study. WOCBP must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]) OR practice abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the patient) from at least 4 weeks prior to first dose to 4 weeks after last dose.

Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or post menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with simultaneous detection of follicle stimulating hormone [FSH] 25 140 IE/L).

Exclusion Criteria:

1. T2DM treated with medication.
2. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
3. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks prior to the first administration of IMP, at the discretion of the Investigator.
4. Any planned major surgery within the duration of the study.
5. Untreated high blood pressure (above 160/100 mmHg at screening).
6. Use of any of the prohibited medication listed in Table 9.6 1 within 2 weeks prior to the first administration of IMP. Recently started use of anti-depressants (e.g., selective serotonin re-uptake inhibitors [SSRI]) within 2 weeks prior to the first IMP administration or planned start of anti-depressant treatment during the study period is not allowed, yet patients that are on stable treatment with anti-depressants for at least two months can be included.
7. Known hypersensitivity to any of the test substances. History of hypersensitivity to drugs with a similar chemical structure or class to orlistat and acarbose.
8. Gastrointestinal problems/diseases, e.g., inflammatory bowel diseases and Irritable Bowel Syndrome (IBS). Untreated gastroesophageal reflux disease (GERD) or GERD that is treated occasionally is allowed as judged by the Investigator.
9. Cholestasis.
10. Previous gastrointestinal surgery that might influence gastrointestinal function significantly, previous bariatric surgery, and previous gallbladder surgery as judged by the investigator.
11. Known vitamin B12 deficiency or other signs of achlorhydria.
12. Chronical malabsorption syndrome.
13. Clinically significant abnormal laboratory values at screening as judged by the investigator.
14. History of severe allergic, cardiac or hepatic disease. History of significant cardiovascular disease such as myocardial infarction, congestive heart failure, stroke, serious cardiac arrhythmias. History of angina within 6 months prior to screening.
15. A personal or family history of Medullary Thyroid Carcinoma (MTC).
16. A personal or family history of Multiple Endocrine Neoplasia syndrome type 2 (MEN 2).
17. Current or history of alcohol abuse and/or use of anabolic steroids or drugs of abuse, as judged by the Investigator.
18. Positive screen for drugs of abuse at screening or admission to the clinic or positive screen for alcohol at screening or admission to the clinic prior to administration of the IMP.
19. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and HIV.
20. Plasma donation within one month of screening or any blood donation (or corresponding blood loss) during the three months prior to screening.
21. Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or participation in any other clinical study that included drug treatment within three months of the first administration of IMP in this study. Patients consented and screened but not dosed in previous studies are not excluded.
22. Investigator considers the patient unlikely to comply with study procedures, restrictions and requirements.
23. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
24. Prolonged QTcF (>450 ms for males, >470 for females), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
25. Patients with swallowing disorders, which may affect the patient's capability to swallow the IMP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Body weight, relative (%) change from baseline for EMP16-02 (120 mg O/40 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Relative (%) change from baseline in body weight after 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A) as compared to placebo.

SECONDARY OUTCOMES:
Body weight, absolute change from baseline for EMP16-02 (120 mg O/40 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Absolute change from baseline in body weight after 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A) as compared to placebo.
Body weight, relative (%) and absolute change from baseline for EMP16-02 (150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Relative (%) and absolute change from baseline in body weight after 14 and 26 weeks of treatment with EMP16-02 (150 mg O/50 mg A) as compared to placebo.
Proportion of patients with ≥5% and ≥10% decrease in body weight for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Proportion of patients with ≥5% and ≥10% decrease in body weight compared to baseline after 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
BMI, relative (%) and absolute change from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Relative (%) and absolute change from baseline in BMI after 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Waist circumference, absolute change from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Absolute change from baseline in waist circumference after 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Sagittal diameter, absolute change from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Absolute change from baseline in sagittal diameter after 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Percentage body fat, relative (%) and absolute change from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Relative (%) and absolute change from baseline in percentage body fat after 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Questionnaire Satiety and craving, after 14 and 26 weeks for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Questionnaire Satiety and craving (generated by Empros Pharma AB) after 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo, corrected for satiety and craving after standardised breakfast at baseline. The questionnaire is generated by Empros Pharma and consists of 7 questions about sense of hunger, sense of satiety and cravings for certain types of food that needs to be answered on a scale from 0 (not at all) to 9 (extremely much).
Haemoglobin A1C (HbA1c): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting haemoglobin A1C (HbA1c) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Glucose: Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting glucose after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Insulin: Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting insulin after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Total cholesterol: Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting total cholesterol after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
High-density lipoprotein (HDL): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting high-density lipoprotein (HDL) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Low-density lipoprotein (LDL): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting low-density lipoprotein (LDL) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Triglycerides: Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting triglycerides after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Albumin: Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting albumin after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
High-sensitivity C-reactive protein (hs CRP): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting high-sensitivity C-reactive protein (hs CRP) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Alanine aminotransferase (ALT): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting alanine aminotransferase (ALT) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Aspartate aminotransferase (AST): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting aspartate aminotransferase (AST) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Alkaline phosphatase (ALP): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting alkaline phosphatase (ALP) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Gamma-glutamyl transferase (GGT): Relative (%) and absolute change from baseline for EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Relative (%) and absolute change from baseline in fasting gamma-glutamyl transferase (GGT) after 7, 14 and 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Proportion of diabetic (fasting glucose ≥ 7.0 mmol/L) and prediabetic patients (fasting glucose ≥ 6.1 mmol/L and < 7.0 mmol/L) for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Change from baseline in the proportion of diabetic (fasting glucose ≥ 7.0 mmol/L) and prediabetic patients (fasting glucose ≥ 6.1 mmol/L and < 7.0 mmol/L) after 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Blood pressure, relative (%) and absolute change from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 14 and week 26.
  Relative (%) and absolute change from baseline in blood pressure after 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Health and life quality questionnaire (RAND-36), change from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Change from baseline in quality of life after 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo. The questionnaire is owned by RAND Corporation USA and translated to swedish by Registercentrum SydOst (RCSO). The health and quality of life questionnaire consists of 36 questions about how the patient experiences his/her own physical and mental health.
Activity and sleep questionnaire, change from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14 and week 26.
  Change from baseline in activity and sleep after 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo. The questionnaire is generated by Empros Pharma. The activity and sleep questionnaire consists of 2 questions about physical activity and sleep during the previous day/night.
Drop-out rate (overall and GI-related), for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose until the date of drop-out, assessed up to 26 weeks.
  Dropout rate (overall and GI-related) following treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Frequency and severity of AEs, for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose until date of resolution of last AE registered or to End of study visit (week 28), whichever comes first.
  Frequency and severity of AEs during 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Bilirubin (total), clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in bilirubin (total) after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Bilirubin (conjugated), clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in bilirubin (conjugated) after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Calcium, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in calcium after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Creatinine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in creatinine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Phosphate, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in phosphate after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Potassium, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in potassium after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Sodium, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in sodium after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Urea, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in urea after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Haematocrit, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in haematocrit after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Haemoglobin (Hb), clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in haemoglobin (Hb) after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Platelet count, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in platelet count after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Red blood cell (RBC) count, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in Red blood cell (RBC) count after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
White blood cell (WBC) count, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in White blood cell (WBC) count after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Activated Partial Thromboplastin Time (APTT), clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in Activated Partial Thromboplastin Time (APTT) after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Prothrombin Complex International Normalised Ratio (PK[INR]), clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in Prothrombin Complex International Normalised Ratio (PK[INR]) after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Erythrocytes in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in erythrocytes in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Glucose in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in glucose in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Ketones in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in ketones in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Leucocytes in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in leucocytes in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Nitrites in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in nitrites in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
pH in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in pH in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Protein in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in protein in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Specific gravity in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in specific gravity in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Urobilinogen in urine, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in urobilinogen in urine after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
ECG HR interval, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in ECG HR interval after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
ECG PR interval, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in ECG PR interval after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
ECG QRS interval, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in ECG QRS interval after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
ECG QT interval, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in ECG QT interval after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
ECG QTcF interval, clinically significant relative (%) and absolute changes from baseline for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline and week 26.
  Clinically significant relative (%) and absolute changes from baseline in ECG QTcF interval after 26 weeks of treatment with EMP16 02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.
Gastrointestinal symptom rating scale (GSRS), for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, after 2, 4, 6, 8, 14 and 26 weeks.
  GI tolerability after 2, 4, 6, 8, 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.The questionnaire is owned by AstraZeneca. The GSRS consists of 15 questions about gastrointestinal symptoms combined into 5 symtom clusters; reflux, abdominal discomfort, indigestion, constipation and diarrhoea. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
IMP compliance, for EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) | From first dose to last dose (week 26). Measured at baseline, week 7, week 14, and week 26.
  Compliance after 7, 14 and 26 weeks of treatment with EMP16-02 (120 mg O/40 mg A and 150 mg O/50 mg A) as compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Litorp, MD, PhD, Principal Investigator — CTC Clinical Trial Consultants AB; Daniel Wilhelms, MD, PhD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (2):
- Sweden (2):
  - Clinical Trial Consultants AB, Linköping
  - Clinical Trial Consultants AB, Uppsala

IPD SHARING:
Plan to Share IPD: No